CLINICAL TRIAL: NCT00842738
Title: Can Mindfulness Meditation Limit the Progression and/or Increase the Remission of Cervical Dysplasia?
Brief Title: Can Alternative Treatment Have an Impact on Cervical Dysplasia?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: John Brodersen, MD, GP, PhD, Associate Professor, Department and Research Unit of G.P., Institute of Public Health, Uni of Copenhagen
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP05010
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2009-02

CONDITIONS: Cervical Dysplasia
Keywords: Screening; Cervical cancer; Cervical dysplasia; Adverse psychosocial effects; Alternative treatment
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness meditation (Active Comparator): Women with mild dysplasia offered mindfulness meditation
  Interventions: Behavioral: Mindfulness meditation
- No meditation (Other): Women with mild dysplasia offered health care services as usual
  Interventions: Other: No meditation
- Controls (Other): Women with normal cervical cells
  Interventions: Other: Controls

INTERVENTIONS:
Behavioral: Mindfulness meditation — Mindfulness meditation
  Arms: Mindfulness meditation
Other: No meditation — Health care services as usual
  Arms: No meditation
Other: Controls — No intervention
  Arms: Controls

SUMMARY:
In this study two questions will be answered:

* can mindfulness meditation help cell-changed on the cervix to disappear?
* can mindfulness meditation lower the psychological distress when women have abnormal cervical cancer screening results?

DETAILED DESCRIPTION:
200 women, who have participated in cervical cancer screening and have mild dysplasia, will be randomized into two groups; an intervention group and a control group. The intervention group will be asked to do mindfulness meditation twice a week listening to instructions from a CD. 200 additional women having normal cervical screening results will also be included in the project.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 23-29 years
* Participated in cervical cancer screening
* Having mild dysplasia and normal screening results

Exclusion Criteria:

* Women who have previously had dysplasia

Ages: 23 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The degree of cervical dysplasia | 6 months after screening

SECONDARY OUTCOMES:
Psychosocial consequences measured with the COS-CC questionnaire | 1 week, 3 and 9 months after screening

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Research Unit of General Practice, Institute of Public Health, Copenhagen, Denmark